CLINICAL TRIAL: NCT02781103
Title: A Randomized Control, Single Blind, Pilot Study of Electroencephalogram (EEG) and Symptoms After Guided Imagery and Transcranial Direct Current Stimulation (tDCS) in Women With Chronic Pelvic Pain
Brief Title: Guided Imagery and Transcranial Direct Current Stimulation (tDCS) in Women With Chronic Pelvic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Kenneth M Peters, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth M Peters, MD, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-117
Record Dates: First submitted 2016-05-12; First posted 2016-05-24 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Cystitis, Interstitial; Pelvic Pain
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided imagery plus active tDCS (Experimental): Subjects will receive 2 milliamps of electrical stimulation to the brain (transcranial direct stimulation-tDCS) for 20 minutes concurrently while listening to a guided imagery CD specifically designed for women with chronic pelvic pain.
  Interventions: Other: Guided imagery plus active tDCS
- Guided imagery plus Sham tDCS (Sham Comparator): Subjects will receive 2 milliamps of electrical stimulation to the brain (transcranial direct stimulation-tDCS) for only 30 seconds and then the device will be turned off. The device will remain in place, however, for 20 minutes while the subject listens to a guided imagery CD specifically designed for women with chronic pelvic pain.
  Interventions: Other: Guided imagery plus Sham tDCS

INTERVENTIONS:
Other: Guided imagery plus active tDCS — The subject will be positioned in the sitting/reclining position in a quiet room with the lights dimmed. The tDCS device and audio headphones will be placed on the subject's head. The tDCS device to be used is the Soterix Medical 1X1 device using 2.0 mA of current. The electrodes that will be used will be standard sponge electrodes. The subject will listen to a scripted guided imagery CD specifically developed for women with chronic pelvic pain through the audio headphones. The guided imagery plus active tDCS arm will have tDCS for 20 minutes concurrently with Guided Imagery.
  Arms: Guided imagery plus active tDCS
Other: Guided imagery plus Sham tDCS — The subject will be positioned in the sitting/reclining position in a quiet room with the lights dimmed. The tDCS device and audio headphones will be placed on the subject's head. The tDCS device to be used is the Soterix Medical 1X1 device using 2.0 mA of current. The electrodes that will be used will be standard sponge electrodes. The subject will listen to a scripted guided imagery CD specifically developed for women with chronic pelvic pain through the audio headphones. The sham arm will have 30 seconds of tDCS, but after 30 seconds the device will be turned off. The device will remain in place until the subject has listened to 20 minutes of the guided imagery CD.
  Arms: Guided imagery plus Sham tDCS

SUMMARY:
This is a single blind, randomized controlled pilot trial of transcranial direct stimulation (tDCS) intervention or tDCS sham administered with a standardized guided imagery intervention. Up to 25 adult women with chronic pelvic pain will be enrolled and randomized (like a flip of the coin) to achieve a total sample size of 20 women. 10 women in one arm of the study will receive guided imagery with tDCS stimulation. 10 women in the other arm of the study will receive guided imagery with sham tDCS. Subjects will remain blinded until the end of the study.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is a common and often debilitating problem among women. It occurs below the umbilicus and is severe enough to cause functional impairment or require treatment. One of the challenges of treating women with CPP is that a single cause is often lacking. CPP presents as a syndrome of symptoms involving gynecologic, gastrointestinal, urologic, and musculoskeletal symptoms as well as psychosocial conditions such as depression that negatively impact quality of life.

The study will consist of one screening visit that may be divided into two visits if needed to accommodate subject's schedules. The screening visit(s) should take place within four weeks prior to starting the intervention schedule. The following will be completed at the screening visit(s): pelvic/levator exam, body mass index (BMI), last menstrual period, medication use, electroencephalogram (EEG), questionnaires (CAGE-AID Questionnaire, Beck Depression Inventory, Interstitial Cystitis Symptom/Problem Index, Generalized Anxiety Disorder 7 item scale, McGill Pain Questionnaire, Pain Catastrophizing Scale, Visual Analog Scale for pain). The subject will complete 16 intervention visits over 12 weeks.

The study intervention visits will be conducted on the Beaumont Hospital- Royal Oak campus by licensed nurses and/or physicians. The initial 10 sessions will occur Monday through Friday, within a 21-day period (allowing for missed days due to unexpected emergencies and/or inclement weather). Excluding weekends, there should be no more than 2 days between the intervention sessions. Each intervention is 20 minutes in duration. After completing the initial 10 sessions, subjects will complete an additional 6 weekly maintenance sessions according to treatment group.

Objectives:

1. To assess the change in EEG alpha brain waves in women with CPP after guided imagery sessions with tDCS actual or sham treatments.
2. To assess the change in pain, urinary symptoms, and quality of life in women after guided imagery sessions with tDCS actual or sham sessions.

Endpoints:

Primary objective/endpoint: Change in alpha wave frequency on EEG after 10 sessions of tDCS and guided imagery, versus 10 sessions of sham tDCS and guided imagery compared to baseline.

Secondary objective/endpoint:

Change in pain levels (0-10) on a Visual Analog Scale (VAS) after 10 intervention sessions and at end of study compared to baseline.

Hypothesis:

The combination of tDCS and Guided Imagery (GI) will enhance patient outcomes, as evidenced by differences in alpha brain wave changes, pain and quality of life (QOL) measures between tDCS actual and sham treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 to 64 years
* Women must either be unable to become pregnant (are surgically sterile or postmenopausal) or must use an approved method of birth control throughout the study period.
* Self- reported CPP defined as pelvic pain that is non-cyclical and of at least 6 months duration and refractory to other treatments
* Subject agrees to not start any new treatment (medication or otherwise) throughout the study treatment and follow up periods.
* Subject agrees to maintain stable doses of all current medications throughout the study treatment and follow-up period.

Exclusion Criteria:

* Pacemaker
* History of seizures during the last 2 years or diagnosis of epilepsy
* Currently using tobacco
* Parkinson's Disease
* Any condition, including neurological or psychiatric illness, which per investigators' judgement may increase subject risk
* History of Hunner's lesion in the medical record
* Lactation, pregnancy, or refusal to use medically approved/reliable birth control in women of child-bearing potential
* Sacral, pudendal Interstim® or spinal cord stimulator that is "on".
* Contraindications to tDCS stimulation (e.g. metal in the head, implanted brain medical devices, scalp wounds or infections, etc.)
* History of head injury resulting in more than a momentary loss of consciousness during the last 2 years

Note: For the sake of preserving scientific integrity, one or more of the eligibility criteria have been left off the list posted while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Change in alpha wave frequency on EEG | Up to 21 days after the first treatment of tDCS +GI or sham tDCS +GI
  Change in alpha wave frequency on EEG between baseline and up to 21 days after the first treatment of tDCS +GI, versus sham tDCS +GI

SECONDARY OUTCOMES:
Change in pain levels on a 0-10 (no pain to most severe pain) Visual Analog Scale (VAS) | Up to 21 days after the first treatment of tDCS +GI or sham tDCS +GI
  Change in pain levels (0-10) on a Visual Analog Scale (VAS) between baseline and up to 21 days after the first treatment of tDCS +GI, versus sham tDCS +GI

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Beaumont Health
Locations (1):
- Beaumont Hospital-Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No